CLINICAL TRIAL: NCT06563284
Title: HealthcAre sUppoRt fOr Remote HIV pAtients: Use of an App to Support HIV+ Patients to Ensure Continuity of Care and Assess Its Impact on Therapy Adherence and Quality of Life
Brief Title: HealthcAre sUppoRt fOr Remote HIV pAtients
Acronym: AURORA
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera SS. Antonio e Biagio e Cesare Arrigo di Alessandria (Other)
Responsible Party: Sponsor
Other Study IDs: ASO.MInf.22.07
Record Dates: First submitted 2024-08-13; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: HIV Infections
Keywords: HIV/AIDS; Mobile application; Digital Health
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: HIV-infected patients in virological suppression who have been treated with a stable antiretroviral regimen for at least six months
  Interventions: Other: AURORA Mobile App

INTERVENTIONS:
Other: AURORA Mobile App — Enrolled subjects will be asked to download the app for free from their smartphone store.
  Weekly/bi-weekly updates were collected, and therapy adherence was facilitated with timed alerts. Patients completed the EQ-5D-5L, PSQI, PHQ-9 and GAD-7 questionnaires every four months to track quality of life, sleep quality, depression and anxiety.

SUMMARY:
Adherence to antiretroviral therapy (ART) is crucial for treatment success in HIV+ patients. This study proposes the use of a smartphone application, specifically developed for this project, to monitor ART adherence and assess quality of life among HIV+ patients. The aim is to optimize long-term disease management through the early identification of comorbidities and clinical complications

DETAILED DESCRIPTION:
Since the first cases were reported more than 35 years ago, 78 million people have been infected with HIV and 35 million have died from AIDS-related illnesses.

Currently, the availability of TARV regimens associated with good tolerability and high levels of efficacy make it necessary to turn attention toward new standards of efficacy indicative of patients' mental and physical well-being. Indeed, health-related quality of life (HRQoL) is becoming increasingly preponderant as a therapeutic outcome. Despite TARV-related viroimmunologic success, people living with HIV (PLWH) continue to have lower HRQoL than the general population. Indeed, much evidence confirms the impact on quality of life not only of therapeutic treatments but also of social and relationship issues and comorbidities. Improving HRQoL is now, therefore, a primary goal for the care and support of PLWH.

Evaluations of new treatments and interventions to improve care, therefore, require the measurement, in addition to clinical endpoints, of HRQoL using valid and reliable instruments. Therefore, the importance of PROs (Patient Reported Outcomes), which represent the description of the patient's own reported state of health, without any interpretation by clinicians or health care personnel, emerges in this area. In this way, the patient is directly involved in his or her own process of care.

Adherence to TARV is essential for successful treatment and improved quality of life. Unfortunately, non-adherence to treatment is a common problem among HIV-infected patients.

The Covid-19 emergence has significantly revolutionized the health care system leading to the implementation of new modes of care, including the use of technological tools to ensure remote medical care.

The present study, targeting HIV-infected patients undergoing virological suppression, aims to use a smartphone application to facilitate continuity of care remotely, promoting adherence to therapy and thus the effectiveness of TARV, assessing the patient's quality of life and identifying possible comorbidities or other critical clinical

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* HIV-infected patients
* HIV plasma RNA values < 50 copies/mL
* Patients referred to the HIV outpatient clinic at the SC Infectious Diseases of the Azienda Alexandria Hospital
* Patients on a stable antiretroviral regimen for at least 6 months
* Patients who have the ability to download the application under study
* Patients who have signed the informed consent

Exclusion Criteria:

* Newly diagnosed patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected patients in virological suppression who have been treated with a stable antiretroviral regimen for at least six months
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-12-20 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Effective use of the mobile application | 6 months
  Frequency of interaction with the mobile application

SECONDARY OUTCOMES:
Adherence to therapy | Everyday, through study completion (6 months)
  Frequency of click in the mobile application
EuroQol five-dimensional questionnaire | Twice, at baseline and after 4 months
  Quality of life assessment questionnaire
Pittsburgh Sleep Quality index | Twice, at baseline and after 4 months
  Quality of sleep assessment questionnaire
Generalized Anxiety Disorder 7 | Twice, at baseline and after 4 months
  Questionnaire for assessment of generalized anxiety state

CONTACTS AND LOCATIONS:
Locations (1):
- SC Malattie Infettive, Alessandria, Piedmont, Italy